CLINICAL TRIAL: NCT02901483
Title: A Phase 1b/2 Study of PEP503 (Radioenhancer) With Radiotherapy in Combination With Concurrent Chemotherapy for Patients With Head and Neck Cancer
Brief Title: A Study of PEP503 With Radiotherapy in Combination With Concurrent Chemotherapy for Patients With Head and Neck Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: bussiness reason
Sponsor: PharmaEngine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEP503-HN-1002
Record Dates: First submitted 2016-08-31; First posted 2016-09-15 (Estimated); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; Radiotherapy

ARMS (1):
- PEP503+Cisplatin+Radiotheraphy (Experimental): Phase 1b: There are 6 levels (L1- 5% + 40mg/m2 weekly cisplatin, L2- 10% + 40mg/m2 weekly cisplatin, L3- 15% + 40mg/m2 weekly cisplatin, L4-22% + 100mg/m2 tri-weekly cisplatin, L3a- 15% + 100mg/m2 tri-weekly cisplatin, and L5- 33% + 100mg/m2 tri-weekly cisplatin) in this phase 1b study. Only primary tumor will receive PEP503 implementation via intratumor injection. A 3 + 3 dose escalation study design will be adopted in this phase to identify the recommended intratumor injection volumes of PEP503.
  Phase 2: The recommended volume identified from phase 1b will be applied in phase 2 for both primary tumor and ≥ 3 cm lymph node lesions.
  Interventions: Drug: PEP503; Drug: Cisplatin; Radiation: Radiotherapy

INTERVENTIONS:
Drug: PEP503 — PEP503 will be administered by intratumoral route as slow injection
  Other Names: NBTXR3
Drug: Cisplatin — The concurrent chemoradiotherapy. Weekly cisplatin 40 mg/m2 or tri-weekly 100 mg/m2, depending on which dose level patients are in, with a minimum of accumulated 200 mg/m2 during the 7~8 weeks' radiation period.
Radiation: Radiotherapy — Patients will receive 70-72 Gy, 2-2.12 Gy/fraction over 7~8 weeks.

SUMMARY:
It's a prospective, open-label, single arm, nonrandomized study of PEP503 in head and neck squamous cell carcinoma (HNSCC) patients.

* Escalation portion (Phase 1b):A 3 + 3 dose escalation study design will be adopted in this phase to identify the recommended intratumor injection volumes of PEP503.
* Expansion portion (Phase 2): Following confirmation of the recommended volumes, 18 additional patients will be enrolled at the recommended volume level to evaluate for safety and efficacy.

DETAILED DESCRIPTION:
Primary Objectives:

* Phase 1b (dose escalation portion): To assess the safety profile and determine the Dose Limiting Toxicity (DLT) and to define the recommended volumes (doses) of PEP503.
* Phase 2 (expansion portion): To evaluate the anti-tumor activity in terms of the rate of locoregional control at one year and to evaluate the safety profile.

Secondary Objectives:

* Phase 1b: To characterize the body kinetic profile of PEP503.
* Phase 2: Objective tumor response, progression free survival rate at 1 year and pathological response (pR).

The target population is composed by patients who have pathologically confirmed squamous cell carcinoma of oral cavity with disease clinically staged as T4b who are not candidates for surgical resection or T3-4 who decline surgery or medical inoperable, or oropharynx, hypopharynx, or larynx with disease clinical staged as T3-4, without metastasis disease. ECOG performance status 0 or 1 and adequate bone marrow, renal, and hepatic function.

Dose limiting toxicity (DLT) - The DLTs are related to PEP503, injection procedure, or concurrent chemo radiation therapy and occur in the DLT evaluation period. The DLT evaluation period starts from the intratumor injection of PEP503 to 4 weeks after the completion of radiation treatment.

There are 6 levels (Level 1, Level 2, Level 3, Level 4, Level 3a and Level 5) in this phase 1b study. PEP503 will be given at the fixed concentration of 53.3g/L. The starting volume of PEP503 to be injected is 5% (Level 1) of the tumor volume confirmed by MRI.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed squamous cell carcinoma (SCC) of oral cavity, oropharynx, hypopharynx, or larynx
* Locally advanced or recurrent disease of: Oral Cavity:T4b, N any, who are not candidates for surgical resection; or T3-4, N any, who decline surgery or medical inoperable; OR Oropharynx, hypopharynx, or larynx: T3-4, N any
* No evidence of distant metastatic disease, as determined by a negative PET scan or CT scan
* ECOG Performance Status 0 or 1
* Adequate function of bone marrow, kidney and liver:

  * White Blood Cell (WBC) ≥ 3.0 x 109/l
  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/l
  * Platelet count ≥ 100 x 109/l
  * Hemoglobin ≥ 9.0 g/dL
  * Creatinine within normal range, for dose level with tri-weekly cisplatin, estimated GFR ≥ 60 mL/min/1.73m2 or CrCl ≥ mL/min is also required
  * AST ≤ 2.5 x ULN, ALT ≤ 2.5 x ULN and Alkaline phosphatase (ALP) ≤ 2.5 x ULN
  * Bilirubin ≤ 1.5 x ULN
* 20 years of age or older
* All female patients of childbearing potential must have negative urine pregnancy test within 7 days prior to study treatment with PEP503. Fertile patients must agree to use effective contraception during the study

Exclusion Criteria:

* Tumor ulceration combined with vascular risks
* Prior radiotherapy to any area within the planned radiotherapy field
* Uncontrolled intercurrent illness
* Concurrent treatment with any other anticancer therapy
* Participation in any investigational drug study within 4 weeks
* Prior or concurrent non-head and neck malignancies, excluding adequately treated basal or squamous cell cancer of the skin, and in situ cervical cancer, and any other cancer from which the subject has been cancer free for 5 years
* Patients unable to comply with scheduled visits and other study procedures.
* Preexisting neuropathy ≥ Grade 2 (CTCAE)
* Pre-existing hearing impairment > Grade 2 (CTCAE) for patients receiving cisplatin 100 mg/m2
* History of allergic reaction to platinum product

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-10-11 (Actual); Primary Completion 2020-08-17 (Actual); Study Completion 2020-08-17 (Actual)

PRIMARY OUTCOMES:
Phase 1: Determination of the Recommended doses and the Dose Limiting Toxicities (DLT) | 24 months
  To determine the Recommended volumes and the Dose Limiting Toxicities (DLT) of PEP503 administered as intratumor injection, activated by CCRT
Phase 2: The rate of locoregional control at one year | 24 months
  To evaluate the rate of locoregional control at one year after PEP503 intratumor injection
Phase1 and 2: Evaluation of Safety profile of PEP503 | 24 months
  Safety of PEP503, as intratumor injection schedule, activated by CCRT will be assessed in terms of incidence and severity of clinical and laboratory Adverse Events by NCI-CTCAE version 4.0

SECONDARY OUTCOMES:
Phase 1: The body kinetic profile of PEP503 | 24 months
  To characterize the body kinetics on Date of injection(DINJ) of PEP503 administered by intratumor injection before CCRT
Phase 2: Evaluation of objective tumor response as per Response Evaluation Criteria in Solid Tumors (RECIST) | 24 months
  To evaluate the objective tumor rate by using RECIST v1.1 after intratumor injection schedule, activated by CCRT
Phase 2: Pathological response (pR) | 24 months
  If patients receive tumor and/or neck lymph node dissection after treatment, to assess according to the evidence of viable tumor cell
Phase 2: Evalution of progression free survival rate at 1 year | 24 months
  To evaluate the progression free survival rate at 1 year after the intratumor injection of PEP503

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Hsu Wang, M.D., Principal Investigator — Keelung Chang Gung Memeorial Hospital (Lovers Lake Branch)
Locations (1):
- Keelung Chang Gung Memorial Hospital (Lovers Lake Branch), Keelung, Taiwan